CLINICAL TRIAL: NCT06722794
Title: Novel Technique for Fixating the Plate of Ahmed Valve to the Sclera Using a Single Flanged Prolene Suture
Brief Title: Fixating the Plate of Ahmed Valve to the Sclera Using a Flanged Prolene Suture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Collaborators: Magrabi Eye & Ear Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEH-IRB# 310- 1-October-2024; Maghrabi eye hospitals (Other: Maghrabi eye hospitals)
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma
Keywords: Ahmed glaucoma valve, prolene, glaucoma drainage device
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Novel Technique for Fixating the Plate of Ahmed Valve to the Sclera Using a Single Flanged Prolene S (Other): Novel Technique for Fixating the Plate of Ahmed Valve to the Sclera Using a Single Flanged Prolene Suture
  Interventions: Procedure: Novel Technique for Fixating the Plate of Ahmed Valve to the Sclera Using a Single Flanged Prolene Suture

INTERVENTIONS:
Procedure: Novel Technique for Fixating the Plate of Ahmed Valve to the Sclera Using a Single Flanged Prolene Suture — This novel technique of fixating the plate of Ahmed glaucoma valve to the sclera using a single flanged prolene suture is an efficient, safe, fast, and reproducible technique that combines the benefits of both fixing the plate providing excellent stability without the complications of free plate techniques and at the same time, minimizing both the risks of conventional old valve plate fixation techniques and the concerns of the relative technical difficulty of suturing due to the difficult access to the posterior globe

SUMMARY:
this study evaluated new technique for suturing the Ahmed valve device used to treat resistant types of glaucoma

DETAILED DESCRIPTION:
This technique of fixating Ahmed glaucoma valve using flanged prolene suture is an safe, fast, and reproducible technique combines the benefits of fixing the plate with excellent stability with no complications of free plate techniques at the same time, decreasing both the risks of old valve plate fixation techniques and the concerns of the relative technical difficulty

ELIGIBILITY:
Inclusion Criteria:

* Patients with IOP more than 21 mmHg , evidence of progressive optic nerve damage, retinal nerve fiber layer defects or typical glaucomatous visual field defects despite maximal tolerable medical or laser treatment are scheduled for surgery.

Exclusion Criteria:

* The exclusion criteria were as follows: patients below 18 years old, those with active uveitis and angle closure glaucoma patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
long term stability and plate migration | 3 months
  ABSENT MOVEMENT OF THE PLATE WITH NO OTHER COMPLICATIONS

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMIR, MD, Principal Investigator — ZAGAZIG UNIVERSITY AND MAGHRABI EYE HOSPITALS
Locations (1):
- Maghrabi Eye Hospitals, Jeddah, Jedda, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
PERSONAL REASONS